CLINICAL TRIAL: NCT02776449
Title: Pathological Cerebral Venous Drainage System Giving Large Pressure Difference Between Brain and Eye at Upright Posture: a Possible Cause to Normal Tension Glaucoma.
Brief Title: Pressure Difference Between Brain and Eye: a Possible Cause to Normal Tension Glaucoma.
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Västerbotten County Council, Sweden (Other Government)
Responsible Party: Sponsor
Other Study IDs: NTG-ICP_1
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2016-05

CONDITIONS: Normal Tension Glaucoma
MeSH Terms: conditions — Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal Tension Glaucoma: Patients with manifest normal tension glaucoma

SUMMARY:
The main aim of this study is to determine the trans-laminal cribrosa pressure difference (TLCPD) for normal tension glaucoma (NTG) patients from the brain and the eye in supine, upright and minor head down tilt positions. It is also to investigate the venous drainage system in the same body positions.

DETAILED DESCRIPTION:
The trans-lamina cribrosa pressure difference (TLCPD), i.e. the difference between the intraocular pressure (IOP) and the intracranial pressure (ICP) has been suggested as a pathophysiological component in glaucoma. The theory is that high TLCPD, either due to elevated IOP or reduced ICP, can cause glaucomatous damage.

Normal tension glaucoma (NTG) patients has been found to have a slightly reduced ICP when measured in horizontal position. However, in a previous study in healthy adult volunteers the investigators have measured TLCPD at supine, sitting and 9 degree head down tilt positions and found that the TLCPD was posture dependent, with the largest difference in the upright position. Since humans are upright approximately two thirds of the day, one can expect that TLCPD in a diurnal perspective is primarily influenced by the ICP in the upright position.

In this study the TLCPD in different positions in patients with NTG will therefore be measured.

The study will be carried out in three parts.

1. TLCPD will be investigated by simultaneous measurements of IOP and ICP. For IOP the Applanation resonance tonometer (ART), developed by our research group, will be used. ART is independent of gravitation and possible to use in all body postures. In this study measurements will be performed in supine, sitting and head down tilt positions. ICP is measured continuously during the period of body position changes with a CELDA lumbar pressure measurement apparatus.
2. Brain and eye MRI investigation will be performed at a 3 Tesla GE scanner with a new generation 32-channels head coil. The images will be used to measure the cross-section area, the blood flow velocity and the flow direction in the jugular veins, as well as the structural properties of the optic nerve and optic nerve head.
3. Ultrasound imaging, using a high-resolution apparatus, will be performed to study the effects of postural changes on the blood flow velocity and the cross-section area of the right and left internal jugular veins and external jugular veins.

ELIGIBILITY:
Inclusion Criteria:

* Subject has normal tension glaucoma in one or both eyes (glaucomatous optic nerve head and corresponding visual field defects)
* Intraocular pressures before treatment did not exceed 21 mmHg. Occasional measurement up to 24 is accepted.

Exclusion Criteria:

* History of brain disease or brain surgery
* History of other neurologic or ocular disease causing visual field loss
* Use of anticoagulants other than acetylsalicylic acid
* Use of carbonic anhydrase inhibitors
* Previous lumbar puncture
* Claustrophobia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Normal tension glaucoma patients
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Trans-lamina cribrosa pressure difference (TLCPD) | 1 day Single time point measurement
  Difference between intraocular pressure (IOP) and intracranial pressure in different body positions

SECONDARY OUTCOMES:
Postural changes on blood flow velocity and cross-section area of right and left internal jugular veins (IJV) and external jugular veins (EJV) | 1 day Single time point measurement

OTHER OUTCOMES:
Retinal perfusion using 3D Phase contrast magnetic resonance imaging (3DPCMRI) | 1 day Single time point measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jan Malm, MD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Linden C, Qvarlander S, Johannesson G, Johansson E, Ostlund F, Malm J, Eklund A. Normal-Tension Glaucoma Has Normal Intracranial Pressure: A Prospective Study of Intracranial Pressure and Intraocular Pressure in Different Body Positions. Ophthalmology. 2018 Mar;125(3):361-368. doi: 10.1016/j.ophtha.2017.09.022. Epub 2017 Oct 31. PMID 29096996